CLINICAL TRIAL: NCT00118547
Title: Health Behavior Change in Chronic Disease Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Turner, Aaron - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B3319V
Record Dates: First submitted 2005-07-01; First posted 2005-07-11 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Multiple Sclerosis
Keywords: Adherence; Medication; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Behavioral: In home monitoring with feedback

INTERVENTIONS:
Behavioral: In home monitoring with feedback — Behavioral counseling

SUMMARY:
The purpose of this pilot trial is to provide preliminary evidence of the effectiveness of a brief behavioral intervention using telemedicine home monitoring to help individuals with multiple sclerosis adhere to medications that slow disease progression.

DETAILED DESCRIPTION:
There is increasing recognition that coordinated approaches to disease management improve medication adherence. Intervention in chronic illness may be viewed as a multidisciplinary and collaborative process based upon behavioral principles, including the idea that illness management skills are learned and behavior is self-directed, motivation and self-efficacy can affect self care, monitoring and responding to changes in physical and mental health improves adaptation to illness, and the health care system can support or hinder self care. Preliminary findings suggest that telemedicine home monitoring providing cues to medication administration, brief evaluation of potential barriers (e.g., fatigue, cognition, side effects), identification of areas for future education (e.g., additional injection training), and an opportunity for feedback to providers (e.g., side effects) are well tolerated and may improve self monitoring of chronic medical conditions.

The proposed study is a six-month, two group parallel-design, controlled trial to evaluate feasibility and obtain effect size estimates for a behavioral intervention to improve adherence to MS disease modifying therapy (DMT) using telemedicine home monitoring. Monitoring will include brief weekly text-based prompting to complete a series of approximately 10-15 questions regarding factors that are expected to affect adherence to DMT. Areas of assessment will include the development of side effects (e.g., flu-like symptoms), disease specific symptoms (e.g., fatigue), adherence expectation, and DMT self-efficacy. MS clinic staff will examine responses to weekly home monitoring assessment. They will provide telephone follow-up for medical advice, support, specific educational materials, and referral for services if necessary. Potential services will also be informed by Research Project 1, and will follow the general principle that they will be selected from a standardized list (e.g., additional injection training, energy management strategies for fatigue), but tailored to individual patient need based upon information obtained by home monitoring.

Primary outcome measures to assess feasibility will be the percentage of eligible participants who complete the study protocol, and comparisons between home monitoring recipients and controls regarding the overall benefits of participation. Outcomes will be assessed via monthly telephone calls.

ELIGIBILITY:
Inclusion Criteria:

- Must have Multiple Sclerosis and be on a disease modifying therapy

Exclusion Criteria:

- Inability to participate in self-care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
adherence | 3,6 months

CONTACTS AND LOCATIONS:
Overall Officials: Aaron P. Turner, PhD, Principal Investigator — VA Puget Sound Health Care System, Seattle
Locations (1):
- VA Puget Sound Health Care System, Seattle, Seattle, Washington, United States

REFERENCES:
- [Result] Turner AP, Williams RM, Sloan AP, Haselkorn JK. Injection anxiety remains a long-term barrier to medication adherence in multiple sclerosis. Rehabil Psychol. 2009 Feb;54(1):116-21. doi: 10.1037/a0014460. PMID 19618711